CLINICAL TRIAL: NCT07172854
Title: Radikal Prostatektomi Sonrasında Aerobik Egzersiz ve Gevşeme Eğitimlerinin Pelvik Taban Kas Eğitimine İlave Etkileri
Brief Title: Pelvic Floor Muscle Training With Aerobic Exercise and Relaxation After Radical Prostatectomy
Acronym: PFMTinPPUI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ege Nur ATABEY, research asisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-24085; TUBITAK (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-08-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Post Prostatectomy Incontinence; Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: interventions — Exercise; Relaxation Therapy; Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group
  Interventions: Other: Pelvic Floor Muscle Training; Other: Aerobic Exercise; Other: Relaxation Training; Other: Patient Education
- Control Group (Active Comparator): Control Group
  Interventions: Other: Pelvic Floor Muscle Training; Other: Patient Education

INTERVENTIONS:
Other: Pelvic Floor Muscle Training — Supervised PFMT with biofeedback, 3 times per week for 12 weeks, plus home exercises.
Other: Aerobic Exercise — Treadmill walking, moderate intensity (Borg 4-6), 60 minutes/session, 3 times per week for 12 weeks.
  Arms: Intervention Group
Other: Relaxation Training — Guided breathing, imagery, and meditation, once weekly for 12 weeks, in addition to home practice.
  Arms: Intervention Group
Other: Patient Education — Standardized education on urinary incontinence, pelvic anatomy, lifestyle modification, and stress management.

SUMMARY:
Post-prostatectomy urinary incontinence (PP-UI) and erectile dysfunction (ED) are common complications after radical prostatectomy, negatively affecting quality of life. Pelvic floor muscle training (PFMT) is widely recommended as the first-line conservative treatment, but recent evidence suggests that multimodal, structured rehabilitation may further improve recovery.

This randomized controlled trial will investigate the additional effects of aerobic exercise and relaxation training combined with PFMT in men following nerve-sparing robotic-assisted radical prostatectomy. Forty-eight participants aged 40-65 years, within one year post-surgery, who demonstrate voluntary pelvic floor muscle contraction and sufficient cognitive function (MoCA), will be randomly assigned (1:1) to intervention or control groups.

All participants will receive standardized education and a 12-week supervised PFMT program with biofeedback and home-based exercises. The intervention group will additionally perform treadmill-based aerobic exercise three times per week and structured relaxation training once per week.

Primary outcomes include urinary symptoms (ICIQ-MLUTS), erectile function (IIEF-15), and prostate cancer-specific quality of life (EPIC). Secondary outcomes include pad test, ICIQ-SF, 6-minute walk test, MoCA, HADS, and adherence.

This non-commercial study aims to provide high-quality evidence supporting physiotherapy-based multimodal rehabilitation for improved pelvic health and quality of life in men after prostate cancer surgery.

DETAILED DESCRIPTION:
Post-prostatectomy urinary incontinence (PP-UI) and erectile dysfunction (ED) are among the most common and distressing complications following radical prostatectomy (RP), significantly affecting the quality of life and psychosocial well-being of prostate cancer survivors. Although pelvic floor muscle training (PFMT) is widely recommended as the first-line conservative approach to manage these complications, recent evidence highlights the importance of multimodal, structured rehabilitation programs supervised by physiotherapists to optimize continence recovery and sexual function.

This randomized controlled trial aims to investigate the additional effects of aerobic exercise and relaxation training when combined with PFMT in men with urinary incontinence and erectile dysfunction following nerve-sparing robotic-assisted radical prostatectomy. The study is designed as a two-arm parallel-group, single-center trial involving 48 male participants aged between 40 and 65 years. Eligible participants must be within one year post-surgery, demonstrate voluntary pelvic floor muscle contraction, and exhibit sufficient cognitive function as assessed by the Montreal Cognitive Assessment (MoCA).

Participants will be randomly allocated (1:1) into either the intervention group or the control group using a computer-generated block randomization procedure. All participants will receive standardized patient education and a 12-week PFMT protocol guided by biofeedback. The PFMT sessions will be conducted individually by a physiotherapist three times per week and include a home-based exercise program monitored through an exercise diary.

In the intervention group, aerobic exercise and relaxation training will be added to PFMT. Aerobic exercise will consist of treadmill walking at moderate intensity (Modified Borg RPE scale 4-6) for 60 minutes (10 min warm-up, 40 min loading, 10 min cool-down), three times per week for 12 weeks. Relaxation training will be conducted once weekly and will include guided breathing, imagery, and meditation techniques in a quiet, dimly lit environment. Patients will be encouraged to practice these relaxation techniques at home using a standardized script.

Assessments will be performed at baseline and at the end of the 12-week intervention. Primary outcome measures include changes in urinary symptoms (ICIQ-MLUTS), erectile function (IIEF-15), and prostate cancer-specific quality of life (EPIC). Secondary outcomes include objective incontinence severity (1-hour pad test), subjective continence impact (ICIQ-SF), functional exercise capacity (6-minute walk test), cognitive performance (MoCA), psychological status (HADS), and exercise adherence (self-reported exercise diary).

All assessments will be carried out during routine clinical visits. The study does not involve any pharmaceutical or implantable medical products and has no placebo arm. No financial incentives will be provided to participants.

This academic, non-commercial trial is expected to generate high-quality evidence to support the role of multimodal physiotherapy in improving pelvic health outcomes in men following prostate cancer surgery. Findings may guide clinicians and healthcare providers in designing structured, holistic rehabilitation protocols that target both physical and emotional recovery in cancer survivorship.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 40 to 65 years
* Underwent nerve-sparing robotic radical prostatectomy within the past 12 months
* Ability to voluntarily contract pelvic floor muscles
* Cognitive capacity sufficient for cooperation with study assessments and interventions, as determined by the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* Presence of acute illness (e.g., urinary tract infection, respiratory infection, interstitial cystitis, bladder or gastrointestinal bleeding)
* Within the first 3 weeks after prostatectomy surgery (acute postoperative period)
* Neurological disorders or diagnosis of neurogenic bladder
* Diagnosed cognitive or psychiatric disorders
* Preoperative urinary incontinence or erectile dysfunction
* History of prior bladder or prostate surgery before prostatectomy
* Participation in pelvic floor muscle training within the last 6 months
* Refusal to participate or absence of signed informed consent form

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in urinary symptoms | Baseline and at 12 weeks post-intervention
  Assessment of changes in three primary domains:
  Lower urinary tract symptoms will be assessed using the International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms Module (ICIQ-MLUTS). Scores range from 0 to 48, with higher scores indicating more severe urinary symptoms.
  All outcomes will be measured at baseline and at the end of the 12-week intervention period.
Change in Erectile Function (IIEF-15) | Baseline and 12 weeks post-intervention
  Erectile function and sexual health will be assessed using the International Index of Erectile Function (IIEF-15). Scores range from 5 to 75, with higher scores indicating better erectile function.
Change in Prostate Cancer-Specific Quality of Life (EPIC) | Baseline and 12 weeks post-intervention
  Prostate cancer-related quality of life will be measured using the Expanded Prostate Cancer Index Composite (EPIC). Scores range from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) Score | Baseline and 12 weeks
  Cognitive performance will be assessed using the Montreal Cognitive Assessment (MoCA). Scores range from 0 to 30, with higher scores reflecting better cognitive function.
Change in 1-Hour Pad Test Result | Baseline and 12 weeks
  Objective severity of urinary incontinence will be measured using the 1-hour pad test. The pad is weighed before and after the test; higher weight gain indicates more leakage.
Change in ICIQ-Short Form (ICIQ-SF) Score | Baseline and 12 weeks
  The subjective impact of urinary incontinence on daily life will be assessed using the ICIQ-Short Form (ICIQ-SF). Scores range from 0 to 21, with higher scores indicating greater impact and worse continence-related quality of life.
Change in Hospital Anxiety and Depression Scale (HADS) Scores | Baseline and 12 weeks
  Psychological status will be assessed using the Hospital Anxiety and Depression Scale (HADS), which includes anxiety (HADS-A) and depression (HADS-D) subscales. Each subscale ranges from 0 to 21. Higher scores indicate greater emotional distress (worse outcomes).
Change in 6-Minute Walk Test Distance | Baseline and 12 weeks
  Functional exercise capacity will be assessed using the 6-Minute Walk Test (6MWT). The total distance walked in meters will be recorded; greater distance indicates better functional capacity.
Exercise Adherence | Throughout 12-week intervention
  Exercise adherence will be monitored through a self-reported exercise diary. Participants will log completion of home-based pelvic floor, aerobic, and relaxation exercises. Adherence rate will be calculated as a percentage of prescribed sessions completed.